CLINICAL TRIAL: NCT03714009
Title: Effect of Fasting on ICSI Outcomes in Poor Responders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Amira S Dieb, Amira S Dieb, MD, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 88766808
Record Dates: First submitted 2018-09-26; First posted 2018-10-22 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Infertility
Keywords: Infertility; Poor ovarian reserve; Intracytoplasmic sperm injection; fasting
MeSH Terms: conditions — Infertility; Fasting | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting group (Active Comparator): Patients will have periodic fasting for 4 weeks prior to the treatment cycle. The fasting method involves daily fasts of 14-16hours and restrict eating to an 8-10 hour "eating window" as 2-3 or more meals of balanced diet. They should take adequate water and non calorie beverages intake daily (2-3 liters)
  Interventions: Behavioral: Fasting
- Non fasting group (Other): no fasting, patients will have usual balanced diet as 3 meals and 2 snacks all over the day. They should take adequate water and non calorie beverages intake daily (2-3 liters)
  Interventions: Behavioral: No fasting

INTERVENTIONS:
Behavioral: Fasting — Periodic fasting last for 4weeks prior to the treatment cycle. The fasting method involves daily fasts of 14-16hours and restrict eating to an 8-10 hour "eating window" as 2-3 or more meals of balanced diet. Patients should take adequate water and non calorie beverages intake daily (2-3 liters).
  Other Names: Periodic fasting
  Arms: Fasting group
Behavioral: No fasting — Patients will not fast . But they will take balanced food and drink 2 to 3 liters of water and non caloric drinks all the day for 4 weeks
  Arms: Non fasting group

SUMMARY:
This study is a prospective, randomized controlled trial conducted at the In Vitro Fertilization ( IVF) center of the Department of Obstetrics & Gynecology, Kasr El-Ainy Teaching Hospital, Faculty of Medicine, Cairo University, Egypt, from October 2018 to September 2019, to determine the clinical effect of fasting on ICSI outcomes in poor responders 360 participants will be randomized withdrawing closed envelopes for each patient into group A and group B .

Group (A): patients will have periodic fasting for 4 weeks prior to the treatment cycle. The fasting method involves daily fasts of 14-16hours and restrict eating to an 8-10 hour "eating window" as 2-3 or more meals of balanced diet. Group (B): no fasting, patients will have usual balanced diet as 3 meals and 2 snacks all over the day. Both groups should take adequate water and non calorie beverages intake daily (2-3 liters).

All patients will start the ICSI cycle using the same treatment protocol. Primary outcome is clinical pregnancy rate per cycle. Secondary outcomes include Body mass index (BMI) and waist/hip ratio (WHR), fasting insulin , fasting plasma glucose, Homeostatic model assessment (HOMA) index, lipid profile ( Triglycerides (TGs), total cholesterol, High density Lipoprotein (HDL), Low density Lipoprotein (LDL), AntiMullerian Hormone (AMH), Basal Follicle Stimulating Hormone (FSH), Luteinizing Hormone (LH), Estradiol (E2, Days of stimulation , dose of gonadotrophins, number of M II oocytes retrieved, number of grade1and 2 embryos, number of frozen embryos, freeze all cycles, Ovarian Hyperstimulation syndrome (OHSS), Chemical pregnancy rate, clinical pregnancy, twins, abortion, ectopic pregnancy, preterm labour, live birth rate

DETAILED DESCRIPTION:
This study is a prospective, single-blinded (to the outcomes assessor), randomized controlled trial conducted at the In Vitro Fertilization ( IVF) center of the Department of Obstetrics & Gynecology, Kasr El-Ainy Teaching Hospital, Faculty of Medicine, Cairo University, Egypt, from October 2018 to September 2019, to determine the clinical effect of fasting on ICSI outcomes in poor responder patients. Ethical committee approval was obtained. The study will include 360 infertile patients with poor ovarian reserve (POR )diagnosed by low Antral follicle count (AFC)( less than 5 follicles), Elevated basal follicle-stimulating hormone (FSH) (more than 10 IU/mL) and low anti-Mullerian hormone (AMH)(less than 1.5 ng/ml), previous POR (≤three oocytes with a conventional stimulation protocol). Women with diabetes, thyroid disorder or other endocrine dysfunctions, uterine abnormalities were excluded.Also severe oligo-astheno-teratozoospermia or azospermia are excluded.

All patients are informed about the study and consent is given by those who accept to participate.

Careful history taking include infertility type, duration , cause, obstetric history, medical and surgical history and demographic distribution is taken. Full physical examination and 2 dimensional (2D) transvaginal sonography (TVS) are done on day 2 to 5 of menses to assess antral follicle count, uterus and adnexa . Body mass index (BMI) and waist/hip ratio (WHR) are calculated, Blood samples are taken for fasting plasma glucose, lipid profile ( Triglycerides (TGs), total cholesterol, High density Lipoprotein (HDL), Low density Lipoprotein (LDL),AntiMullerian Hormone (AMH), Basal Follicle Stimulating Hormone (FSH), Luteinizing Hormone (LH), Estradiol (E2) All 360 participants will be randomized withdrawing closed envelopes for each patient into group A and group B .

Group (A): patients will have periodic fasting for 4 weeks prior to the treatment cycle. The fasting method involves daily fasts of 14-16hours and restrict eating to an 8-10 hour "eating window" as 2-3 or more meals of balanced diet. Group (B): no fasting, patients will have usual balanced diet as 3 meals and 2 snacks all over the day. Both groups should take adequate water and non calorie beverages intake daily (2-3 liters) Subjects are instructed to wait for spontaneous menses. The next visit is scheduled on day 2 of next cycle when transvaginal ultrasound is done to confirm that endometrial thickness <5mm, no ovarian cyst by ultrasound. Body mass index (BMI) and waist/hip ratio (WHR) are calculated. Blood samples are taken for fasting plasma glucose, lipid profile ( Triglycerides (TGs), total cholesterol, High density Lipoprotein (HDL), Low density Lipoprotein (LDL), AntiMullerian Hormone (AMH), Basal Follicle Stimulating Hormone (FSH), Luteinizing Hormone (LH), Estradiol (E2),and then antagonist protocol is followed. Gonadotropins as Intramuscular (I.M.) injections of 150-300 (International units) I.U. of highly purified Human Menopausal Gonadotropins daily (Merional, 75 I.U. /vial, IBSA). and Urofollitropin or highly purified human follicle stimulating hormone(Fostimon®, 75 I.U. /vial, IBSA) are give in a ratio of 1:1.The dose is adjusted according to the age, BMI, Antral follicle count (AFC), serum levels of AMH, FSH and ovarian response.

On the sixth day of stimulation , a visit is scheduled to assess the ovarian response ( folliculometry) by TVS. Gonadotrophin releasing hormone antagonist (GnRH antagonist) which is Cetrorelix 0.25mg ( Cetrotide®, 0.25 mg/ vial, Merck Serono, is filled and mixed with diluent from a prefilled syringe with a 20 gauge needle) is given subcutaneously (S.C.) by 27-gauge needle starting from the 6th day of stimulation (fixed antagonist protocol).

Next visits are every other day for follow up using the TVS. The trigger by Human Chorionic Gonadotrophin (HCG)10000 I.U., I.M. ( Pregnyl, Organon) is given when at least 3 follicles reach 18mm in mean diameter or more and E2 level is less than 2500 pg/ml. Ovum retrieval is done 34 hours after HCG injection and embryo transfer using Wallace catheter on day 2 to 3. Luteal support includes natural Progesterone 400 mg 1x2 as rectal suppository, Folic acid 0.5 mg orally once daily, Amoxicillin-Clavulanic Acid 1gm 1x2x7 orally, Progesterone 100 I.M. injections daily for 10 days, Acetylsalicylic Acid (75 mg) orally once daily Quantitative ß- HCG in serum after is done after 14 days of embryo transfer.TVS is performed to detect clinical pregnancy at 6-7 weeks of gestation.

Primary outcome is clinical pregnancy rate per cycle. Secondary outcomes include Body mass index (BMI) and waist/hip ratio (WHR), fasting plasma glucose, lipid profile ( Triglycerides (TGs), total cholesterol, High density Lipoprotein (HDL), Low density Lipoprotein (LDL), AntiMullerian Hormone (AMH), Basal Follicle Stimulating Hormone (FSH), Luteinizing Hormone (LH), Estradiol (E2, Days of stimulation , dose of gonadotrophins, number of M II oocytes retrieved, number of grade1and 2 embryos, number of frozen embryos, freeze all cycles, Ovarian Hyperstimulation syndrome (OHSS), Chemical pregnancy rate, clinical pregnancy, twins, abortion, ectopic pregnancy, preterm labour, live birth rate

ELIGIBILITY:
The study will include:

infertile patients with poor ovarian reserve (POR )diagnosed by low Antral follicle count (AFC)( less than 5 follicles), Elevated basal follicle-stimulating hormone (FSH) (more than 10 IU/mL) and low anti-Mullerian hormone (AMH)(less than 1.5 ng/ml), previous POR (≤three oocytes with a conventional stimulation protocol).

Women with diabetes, thyroid disorder or other endocrine dysfunctions, uterine abnormalities were excluded.Also severe oligo-astheno-teratozoospermia or azospermia are excluded.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 360 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate per cycle | 10 weeks
  detection of gestationalsac, embryonal pole and fetal pulsations by ultrasonography

SECONDARY OUTCOMES:
Body mass index | 4 weeks of fasting
  The weight in kilograms divided by the squared height in meters
Waist/Hip ratio | 4 weeks of fasting
  The ratio of waist circumference in centimeters to the hip circumference in centimeters
Number of days of stimulation with gonadotrophins | 6 weeks
  Days of stimulation with gonadotrophins
Number of ampoules of gonadotrophins | 6 weeks
  total number of ampoules of gonadotrophins
number of M II oocytes retrieved | 6 weeks
  number of M II oocytes retrieved
number of grade1and 2 embryos | 6-7 weeks
  number of grade1and 2 embryos
number of frozen embryos | 6-7 weeks
  number of frozen embryos
number of freeze all cycles | 6 weeks
  total number of freeze all cycles
number of cancelled cycles | 6 weeks
  total number of cancelled cycles
Rate of chemical pregnancy rate | 10 weeks
  number of cases with positive pregnancy test with no clinical pregnancy
Rate of twin pregnancy | 10 weeks
  presence of two gestational sacs detected by ultrasonography
Rate of abortion per cycle | 10-24 weeks after embryo transfer
  number of abortions clinically detected per cycle
Rate of ectopic pregnancy | 10 weeks
  the presence of gestational sac outside the uterine cavity detected by ultrasound
Rate of preterm labour | After 24 weeks of start of study
  labour after 20 weeks of gestation and before completed 37 weeks of gestation
live birth rate | After40 weeks of start of study
  live birth rate

CONTACTS AND LOCATIONS:
Overall Officials: Amira S Dieb, MD, Principal Investigator — KasrAlainiH
Locations (1):
- KasrELAiniH, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No